CLINICAL TRIAL: NCT04278755
Title: A Mechanistic Examination of Continuous Cycle Oral Contractive Administration in Binge Eating
Brief Title: Binge Eating & Birth Control
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted prematurely due to COVID-19-related enrollment challenges.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-3149
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-06

CONDITIONS: Bulimia Nervosa; Binge Eating; Eating Disorders; Binge-Eating Disorder
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Feeding and Eating Disorders; Binge-Eating Disorder | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Continuous OC (Experimental): Continuous daily oral drospirenone + ethinyl estradiol for 84 days (i.e., 12-weeks).
  Interventions: Drug: Drospirenone-Ethinyl Estradiol Oral Tablet

INTERVENTIONS:
Drug: Drospirenone-Ethinyl Estradiol Oral Tablet — 3 Mg-0.03 Mg continuous daily Drospirenone-Ethinyl Estradiol.
  Other Names: Yasmin

SUMMARY:
This pilot study examines the effect of stabilizing ovarian hormones on eating behaviors and brain activation in women with binge eating (n=15) using functional magnetic resonance imaging (fMRI) and behavioral tests. This is completed by taking oral contraceptives (birth control) continuously for three months. Prior to medication administration and at the end of treatment, eating behaviors will be measured and fMRI will be conducted in order to examine changes in activation in dopamine-reward pathways that occur with oral contraceptive administration. This will assess changes in brain activation that occur with the stabilization of ovarian hormones.

DETAILED DESCRIPTION:
Eating disorders (EDs) affect 15 million women in the United States and have one of the highest mortality rates of any mental illness. Despite this, the underlying neurobiology remains poorly understood. EDs predominantly occur in women, and the frequency of certain symptoms change in a predictable pattern over the menstrual cycle; specifically, symptom changes appear to be triggered by normal fluctuations in the ovarian hormones estradiol (E2) and progesterone (P4).

The objective of this study is to examine the impact of ovarian hormone stabilization, through the continuous administration of oral contraceptives (OCs) for 3-months, on brain activation in response to reward and eating behaviors in women who binge eat (n=15) using functional magnetic resonance imaging (fMRI) and behavioral testing. OCs work by suppressing ovulation, thereby reducing E2 and P4 changes that occur pre- and post- ovulation. Because the traditional 21/7 regimen of OC administration (21 active pills followed by 7 days of inactive pills) allows follicles to begin to develop, this leads to the secretion of endogenous E2, and then E2 withdrawal once active pills begin again. This does not result in consistent stabilization. Thus, this study will use OCs in a continuous manner, with no inactive pills.

Participants will complete fMRI imaging and self-report questionnaires prior to OC administration and at the end of OC administration. The investigators will examine within-subject changes that occur in these measures with OC administration. The primary hypothesis is that continuous OC treatment will have a beneficial/stabilizing effect on outcomes of interest. Specifically, symptomatology may decrease from OC use. Results will ultimately provide the pilot data necessary for larger mechanistic trials.

The specific aims are to:

Aim 1: Quantify the effect of ovarian hormone stabilization on eating behaviors in women with binge eating.

Aim 2: Examine the effect of ovarian hormone stabilization on response to reward using fMRI and self-report questionnaires in women with binge eating.

ELIGIBILITY:
Inclusion Criteria

Participants will include women ages 18-34 with a current Diagnostic and Statistical Manual (DSM-5) diagnosis of a binge eating syndrome and a regular menstrual cycle. Only participants capable of giving informed consent and understanding the risks associated with the study will be enrolled.

* Current binge eating behaviors meeting DSM-5 criteria for a binge eating syndrome
* Age 18-34
* Regular menstrual cycle for at least 3-months
* Free of medication or medical condition that impacts ovarian hormones or is contraindicated for use with study interventions (including birth control)
* Speaks English

Exclusion Criteria

* any foreign metal objects or implants in your body as determined by the safety questionnaires (due to fMRI)
* use of birth control or hormones in the past 3-months
* hormonal contraceptives that are implanted (i.e. progestin intrauterine device or implant)
* current pregnancy, lactation, or < 12-weeks postpartum
* previous serious, negative reaction to birth control
* current smoker
* < 18.5 BMI > 31
* history of bipolar disorder or psychotic episodes
* frequent laxative and/or diuretic use
* previous suicide attempt
* abnormal/undiagnosed vaginal bleeding; endometriosis
* recurrent migraine headaches or headaches with focal neurological symptoms
* hypertension or vascular disease (i.e., coronary artery disease, congestive heart failure, cerebrovascular disease)
* diabetes or other circulation problems
* blood clotting disorder
* porphyria
* breast, uterus/cervix, or vaginal cancer
* medical condition or medication use that increases serum potassium levels (including frequent laxative or diuretic use)
* high cholesterol
* history of venous thromboembolus (VTE), deep vein thrombosis, pulmonary embolism, phlebothrombosis, coronary thrombosis, thromboembolism, thrombophlebitis, or any type of blood clot or blood clot disorder (e.g., thromboembolic disease, Factor V Leiden), protein C or S deficiency, heart attack or stroke, atrial fibrillation, heart, liver, kidney, or adrenal disease, endocarditis, liver cancer, malignant melanoma, cholecystitis or pancreatitis, VTE or jaundice caused by pregnancy or birth control pills, recent significant period of immobility (e.g., pregnancy bed rest), immediate family history of a hereditary blood clotting disorder
* Pregnant women will be excluded from participation and women who become pregnant (although unlikely) will be withdrawn. Prior to enrollment, a pregnancy test will be completed. All participants will be required to use non-hormonal forms of birth control (e.g., barrier methods) to avoid pregnancy during this study. If a woman becomes pregnant during the study, participation will be discontinued.
* Any condition or symptoms considered by the study team to detrimentally impact subject safety.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Men will not be included in this study given the stated purpose to study ovarian hormones.
Enrollment: 8 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Baker, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 18 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with University of North Carolina (UNC).
Supporting Information: SAP, Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 18 to 24 months following publication upon reasonable request.
Access Criteria: Approval from an IRB, IEC, or REB, as applicable and execution of a data use/sharing agreement with UNC.

REFERENCES:
- [Background] American Psychiatric Association, Diagnostic and Statistical Manual of Mental Disorders. Fifth Edition. 2013, Washington, DC: American Psychiatric Press.
- [Background] Baker JH, Girdler SS, Bulik CM. The role of reproductive hormones in the development and maintenance of eating disorders. Expert Rev Obstet Gynecol. 2012 Nov 1;7(6):573-583. doi: 10.1586/eog.12.54. PMID 23585773
- [Background] Edler C, Lipson SF, Keel PK. Ovarian hormones and binge eating in bulimia nervosa. Psychol Med. 2007 Jan;37(1):131-41. doi: 10.1017/S0033291706008956. Epub 2006 Oct 12. PMID 17038206
- [Background] Lester NA, Keel PK, Lipson SF. Symptom fluctuation in bulimia nervosa: relation to menstrual-cycle phase and cortisol levels. Psychol Med. 2003 Jan;33(1):51-60. doi: 10.1017/s0033291702006815. PMID 12537036
- [Background] Price WA, Torem MS, DiMarzio LR. Premenstrual exacerbation of bulimia. Psychosomatics. 1987 Jul;28(7):378-9. doi: 10.1016/s0033-3182(87)72511-0. No abstract available. PMID 3438453
- [Background] Gladis MM, Walsh BT. Premenstrual exacerbation of binge eating in bulimia. Am J Psychiatry. 1987 Dec;144(12):1592-5. doi: 10.1176/ajp.144.12.1592. PMID 3688285
- [Background] Asarian L, Geary N. Modulation of appetite by gonadal steroid hormones. Philos Trans R Soc Lond B Biol Sci. 2006 Jul 29;361(1471):1251-63. doi: 10.1098/rstb.2006.1860. PMID 16815802
- [Background] Naessen S, Carlstrom K, Bystrom B, Pierre Y, Hirschberg AL. Effects of an antiandrogenic oral contraceptive on appetite and eating behavior in bulimic women. Psychoneuroendocrinology. 2007 Jun;32(5):548-54. doi: 10.1016/j.psyneuen.2007.03.008. Epub 2007 May 2. PMID 17475412
- [Background] Monteleone AM, Monteleone P, Esposito F, Prinster A, Volpe U, Cantone E, Pellegrino F, Canna A, Milano W, Aiello M, Di Salle F, Maj M. Altered processing of rewarding and aversive basic taste stimuli in symptomatic women with anorexia nervosa and bulimia nervosa: An fMRI study. J Psychiatr Res. 2017 Jul;90:94-101. doi: 10.1016/j.jpsychires.2017.02.013. Epub 2017 Feb 21. PMID 28249187
- [Background] Forbush KT, Wildes JE, Pollack LO, Dunbar D, Luo J, Patterson K, Petruzzi L, Pollpeter M, Miller H, Stone A, Bright A, Watson D. Development and validation of the Eating Pathology Symptoms Inventory (EPSI). Psychol Assess. 2013 Sep;25(3):859-78. doi: 10.1037/a0032639. Epub 2013 Jul 1. PMID 23815116
- [Background] Franken IH, Muris P, Georgieva I. Gray's model of personality and addiction. Addict Behav. 2006 Mar;31(3):399-403. doi: 10.1016/j.addbeh.2005.05.022. Epub 2005 Jun 16. PMID 15964149
- [Background] Harrison A, O'Brien N, Lopez C, Treasure J. Sensitivity to reward and punishment in eating disorders. Psychiatry Res. 2010 May 15;177(1-2):1-11. doi: 10.1016/j.psychres.2009.06.010. Epub 2010 Apr 9. PMID 20381877
- [Background] Knutson B, Westdorp A, Kaiser E, Hommer D. FMRI visualization of brain activity during a monetary incentive delay task. Neuroimage. 2000 Jul;12(1):20-7. doi: 10.1006/nimg.2000.0593. PMID 10875899
- [Background] Le Strat Y, Dubertret C, Le Foll B. Prevalence and correlates of major depressive episode in pregnant and postpartum women in the United States. J Affect Disord. 2011 Dec;135(1-3):128-38. doi: 10.1016/j.jad.2011.07.004. Epub 2011 Jul 29. PMID 21802737
- [Background] Lee EE, Nieman LK, Martinez PE, Harsh VL, Rubinow DR, Schmidt PJ. ACTH and cortisol response to Dex/CRH testing in women with and without premenstrual dysphoria during GnRH agonist-induced hypogonadism and ovarian steroid replacement. J Clin Endocrinol Metab. 2012 Jun;97(6):1887-96. doi: 10.1210/jc.2011-3451. Epub 2012 Mar 30. PMID 22466349
- [Background] Legro RS, Ary BA, Paulson RJ, Stanczyk FZ, Sauer MV. Premature luteinization as detected by elevated serum progesterone is associated with a higher pregnancy rate in donor oocyte in-vitro fertilization. Hum Reprod. 1993 Sep;8(9):1506-11. doi: 10.1093/oxfordjournals.humrep.a138288. PMID 8253943
- [Background] Leibenluft E, Schmidt PJ, Turner EH, Danaceau MA, Ashman SB, Wehr TA, Rubinow DR. Effects of leuprolide-induced hypogonadism and testosterone replacement on sleep, melatonin, and prolactin secretion in men. J Clin Endocrinol Metab. 1997 Oct;82(10):3203-7. doi: 10.1210/jcem.82.10.4270. PMID 9329339
- [Background] Leibenluft E. Pediatric Irritability: A Systems Neuroscience Approach. Trends Cogn Sci. 2017 Apr;21(4):277-289. doi: 10.1016/j.tics.2017.02.002. Epub 2017 Mar 6. PMID 28274677
- [Background] Leibenluft E, Cohen P, Gorrindo T, Brook JS, Pine DS. Chronic versus episodic irritability in youth: a community-based, longitudinal study of clinical and diagnostic associations. J Child Adolesc Psychopharmacol. 2006 Aug;16(4):456-66. doi: 10.1089/cap.2006.16.456. PMID 16958570
- [Background] Li CI, Malone KE, Porter PL, Weiss NS, Tang MT, Cushing-Haugen KL, Daling JR. Relationship between long durations and different regimens of hormone therapy and risk of breast cancer. JAMA. 2003 Jun 25;289(24):3254-63. doi: 10.1001/jama.289.24.3254. PMID 12824206
- [Background] Licciardi F, Berkeley AS, Krey L, Grifo J, Noyes N. A two- versus three-embryo transfer: the oocyte donation model. Fertil Steril. 2001 Mar;75(3):510-3. doi: 10.1016/s0015-0282(00)01755-6. PMID 11239533
- [Background] Licciardi FL, Kwiatkowski A, Noyes NL, Berkeley AS, Krey LL, Grifo JA. Oral versus intramuscular progesterone for in vitro fertilization: a prospective randomized study. Fertil Steril. 1999 Apr;71(4):614-8. doi: 10.1016/s0015-0282(98)00515-9. PMID 10202868
- [Background] Lobo RA. Evaluation of cardiovascular event rates with hormone therapy in healthy, early postmenopausal women: results from 2 large clinical trials. Arch Intern Med. 2004 Mar 8;164(5):482-4. doi: 10.1001/archinte.164.5.482. No abstract available. PMID 15006823
- [Background] Lopez OL, Becker JT, Sweet RA, Klunk W, Kaufer DI, Saxton J, Habeych M, DeKosky ST. Psychiatric symptoms vary with the severity of dementia in probable Alzheimer's disease. J Neuropsychiatry Clin Neurosci. 2003 Summer;15(3):346-53. doi: 10.1176/jnp.15.3.346. PMID 12928511
- [Background] Lukaszuk K, Liss J, Lukaszuk M, Maj B. Optimization of estradiol supplementation during the luteal phase improves the pregnancy rate in women undergoing in vitro fertilization-embryo transfer cycles. Fertil Steril. 2005 May;83(5):1372-6. doi: 10.1016/j.fertnstert.2004.11.055. PMID 15866571
- [Background] Mandel FP, Geola FL, Meldrum DR, Lu JH, Eggena P, Sambhi MP, Hershman JM, Judd HL. Biological effects of various doses of vaginally administered conjugated equine estrogens in postmenopausal women. J Clin Endocrinol Metab. 1983 Jul;57(1):133-9. doi: 10.1210/jcem-57-1-133. PMID 6304131
- [Background] Manson JE, Hsia J, Johnson KC, Rossouw JE, Assaf AR, Lasser NL, Trevisan M, Black HR, Heckbert SR, Detrano R, Strickland OL, Wong ND, Crouse JR, Stein E, Cushman M; Women's Health Initiative Investigators. Estrogen plus progestin and the risk of coronary heart disease. N Engl J Med. 2003 Aug 7;349(6):523-34. doi: 10.1056/NEJMoa030808. PMID 12904517
- [Background] Matthews KA, Berga SL, Owens JF, Flory JD. Effects of short-term suppression of ovarian hormones on cardiovascular and neuroendocrine reactivity to stress in women. Psychoneuroendocrinology. 1998 May;23(4):307-22. doi: 10.1016/s0306-4530(98)00013-4. PMID 9695133
- [Background] McGuire K, Fung LK, Hagopian L, Vasa RA, Mahajan R, Bernal P, Silberman AE, Wolfe A, Coury DL, Hardan AY, Veenstra-VanderWeele J, Whitaker AH. Irritability and Problem Behavior in Autism Spectrum Disorder: A Practice Pathway for Pediatric Primary Care. Pediatrics. 2016 Feb;137 Suppl 2:S136-48. doi: 10.1542/peds.2015-2851L. Epub 2016 Feb 1. PMID 26908469
- [Background] McLaren DG, Ries ML, Xu G, Johnson SC. A generalized form of context-dependent psychophysiological interactions (gPPI): a comparison to standard approaches. Neuroimage. 2012 Jul 16;61(4):1277-86. doi: 10.1016/j.neuroimage.2012.03.068. Epub 2012 Mar 30. PMID 22484411
- [Background] McNaughton N, Corr PJ. A two-dimensional neuropsychology of defense: fear/anxiety and defensive distance. Neurosci Biobehav Rev. 2004 May;28(3):285-305. doi: 10.1016/j.neubiorev.2004.03.005. PMID 15225972
- [Background] Melis GB, Fruzzetti F, Paoletti AM, Carmassi F, Fioretti P. Fibrinopeptide A plasma levels during low-estrogen oral contraceptive treatment. Contraception. 1984 Dec;30(6):575-83. doi: 10.1016/0010-7824(84)90007-6. PMID 6241562
- [Background] Mezrow G, Shoupe D, Spicer D, Lobo R, Leung B, Pike M. Depot leuprolide acetate with estrogen and progestin add-back for long-term treatment of premenstrual syndrome. Fertil Steril. 1994 Nov;62(5):932-7. PMID 7926137
- [Background] Mirkin S, Gimeno TG, Bovea C, Stadtmauer L, Gibbons WE, Oehninger S. Factors associated with an optimal pregnancy outcome in an oocyte donation program. J Assist Reprod Genet. 2003 Oct;20(10):400-8. doi: 10.1023/a:1026236726568. PMID 14649379
- [Background] Mitwally MF, Gotlieb L, Casper RF. Prevention of bone loss and hypoestrogenic symptoms by estrogen and interrupted progestogen add-back in long-term GnRH-agonist down-regulated patients with endometriosis and premenstrual syndrome. Menopause. 2002 Jul-Aug;9(4):236-41. doi: 10.1097/00042192-200207000-00004. PMID 12082359
- [Background] Mogg K, Bradley BP. Some methodological issues in assessing attentional biases for threatening faces in anxiety: a replication study using a modified version of the probe detection task. Behav Res Ther. 1999 Jun;37(6):595-604. doi: 10.1016/s0005-7967(98)00158-2. PMID 10372472
- [Background] Mogg, K., & Bradley, B. P. (2005). Attentional Bias in Generalized Anxiety Disorder Versus Depressive Disorder. Cognitive Therapy and Research, 29(1), 29-45. https://doi.org/10.1007/s10608-005-1646-y
- [Background] Moses-Kolko EL, Fraser D, Wisner KL, James JA, Saul AT, Fiez JA, Phillips ML. Rapid habituation of ventral striatal response to reward receipt in postpartum depression. Biol Psychiatry. 2011 Aug 15;70(4):395-9. doi: 10.1016/j.biopsych.2011.02.021. Epub 2011 Apr 20. PMID 21507385
- [Background] Moses-Kolko EL, Perlman SB, Wisner KL, James J, Saul AT, Phillips ML. Abnormally reduced dorsomedial prefrontal cortical activity and effective connectivity with amygdala in response to negative emotional faces in postpartum depression. Am J Psychiatry. 2010 Nov;167(11):1373-80. doi: 10.1176/appi.ajp.2010.09081235. Epub 2010 Sep 15. PMID 20843875
- [Background] Murphy KJ, Brunberg JA. Adult claustrophobia, anxiety and sedation in MRI. Magn Reson Imaging. 1997;15(1):51-4. doi: 10.1016/s0730-725x(96)00351-7. PMID 9084025
- [Background] Nagy ZP, Chang CC, Shapiro DB, Bernal DP, Elsner CW, Mitchell-Leef D, Toledo AA, Kort HI. Clinical evaluation of the efficiency of an oocyte donation program using egg cryo-banking. Fertil Steril. 2009 Aug;92(2):520-6. doi: 10.1016/j.fertnstert.2008.06.005. Epub 2008 Aug 9. PMID 18692830
- [Background] Nieman, L. K., & Loriaux, D. L. (1992). Estrogens and progestins. In Textbook of pharmacology (pp. 695-716). Philadelphia, PA: W.B. Saunders Company.
- [Background] Noyes N, Hampton BS, Berkeley A, Licciardi F, Grifo J, Krey L. Factors useful in predicting the success of oocyte donation: a 3-year retrospective analysis. Fertil Steril. 2001 Jul;76(1):92-7. doi: 10.1016/s0015-0282(01)01823-4. PMID 11438325
- [Background] Oates M. Perinatal psychiatric disorders: a leading cause of maternal morbidity and mortality. Br Med Bull. 2003;67:219-29. doi: 10.1093/bmb/ldg011. PMID 14711766
- [Background] Padilla SL, Smith RD, Garcia JE. The Lupron screening test: tailoring the use of leuprolide acetate in ovarian stimulation for in vitro fertilization. Fertil Steril. 1991 Jul;56(1):79-83. doi: 10.1016/s0015-0282(16)54421-5. PMID 1906020
- [Background] Paulson RJ, Hatch IE, Lobo RA, Sauer MV. Cumulative conception and live birth rates after oocyte donation: implications regarding endometrial receptivity. Hum Reprod. 1997 Apr;12(4):835-9. doi: 10.1093/humrep/12.4.835. PMID 9159452
- [Background] Penn DL, Spaulding W, Reed D, Sullivan M. The relationship of social cognition to ward behavior in chronic schizophrenia. Schizophr Res. 1996 Jul 5;20(3):327-35. doi: 10.1016/0920-9964(96)00010-2. PMID 8827860
- [Background] Peress MR, Phillips HM. Quintuplet gestation following transfer of five cryopreserved embryos: conditions stimulating thawed-embryo implantation. J Assist Reprod Genet. 1998 Sep;15(8):521-3. doi: 10.1023/a:1022590605998. No abstract available. PMID 9785200
- [Background] Perlis RH, Fraguas R, Fava M, Trivedi MH, Luther JF, Wisniewski SR, Rush AJ. Prevalence and clinical correlates of irritability in major depressive disorder: a preliminary report from the Sequenced Treatment Alternatives to Relieve Depression study. J Clin Psychiatry. 2005 Feb;66(2):159-66; quiz 147, 273-4. PMID 15705000
- [Background] Petitti DB, Sidney S, Perlman JA. Increased risk of cholecystectomy in users of supplemental estrogen. Gastroenterology. 1988 Jan;94(1):91-5. doi: 10.1016/0016-5085(88)90614-2. PMID 3335303
- [Background] Pizzagalli DA, Holmes AJ, Dillon DG, Goetz EL, Birk JL, Bogdan R, Dougherty DD, Iosifescu DV, Rauch SL, Fava M. Reduced caudate and nucleus accumbens response to rewards in unmedicated individuals with major depressive disorder. Am J Psychiatry. 2009 Jun;166(6):702-10. doi: 10.1176/appi.ajp.2008.08081201. Epub 2009 May 1. PMID 19411368
- [Background] Postpartum Depression: Action Towards Causes and Treatment (PACT) Consortium. Heterogeneity of postpartum depression: a latent class analysis. Lancet Psychiatry. 2015 Jan;2(1):59-67. doi: 10.1016/S2215-0366(14)00055-8. Epub 2015 Jan 8. PMID 26359613
- [Background] Prentice RL, Langer RD, Stefanick ML, Howard BV, Pettinger M, Anderson GL, Barad D, Curb JD, Kotchen J, Kuller L, Limacher M, Wactawski-Wende J; Women's Health Initiative Investigators. Combined analysis of Women's Health Initiative observational and clinical trial data on postmenopausal hormone treatment and cardiovascular disease. Am J Epidemiol. 2006 Apr 1;163(7):589-99. doi: 10.1093/aje/kwj079. Epub 2006 Feb 16. PMID 16484450
- [Background] Prentice RL, Langer R, Stefanick ML, Howard BV, Pettinger M, Anderson G, Barad D, Curb JD, Kotchen J, Kuller L, Limacher M, Wactawski-Wende J; Women's Health Initiative Investigators. Combined postmenopausal hormone therapy and cardiovascular disease: toward resolving the discrepancy between observational studies and the Women's Health Initiative clinical trial. Am J Epidemiol. 2005 Sep 1;162(5):404-14. doi: 10.1093/aje/kwi223. Epub 2005 Jul 20. PMID 16033876
- [Background] Price M, van Stolk-Cooke K. Examination of the interrelations between the factors of PTSD, major depression, and generalized anxiety disorder in a heterogeneous trauma-exposed sample using DSM 5 criteria. J Affect Disord. 2015 Nov 1;186:149-55. doi: 10.1016/j.jad.2015.06.012. Epub 2015 Jul 29. PMID 26241663
- [Background] Rice VC, Richard-Davis G, Saleh AA, Ginsburg KA, Mammen EF, Moghissi K, Leach R. Fibrinolytic parameters in women undergoing ovulation induction. Am J Obstet Gynecol. 1993 Dec;169(6):1549-53. doi: 10.1016/0002-9378(93)90434-k. PMID 8267060
- [Background] Rich BA, Holroyd T, Carver FW, Onelio LM, Mendoza JK, Cornwell BR, Fox NA, Pine DS, Coppola R, Leibenluft E. A preliminary study of the neural mechanisms of frustration in pediatric bipolar disorder using magnetoencephalography. Depress Anxiety. 2010 Mar;27(3):276-86. doi: 10.1002/da.20649. PMID 20037920
- [Background] Rich BA, Schmajuk M, Perez-Edgar KE, Fox NA, Pine DS, Leibenluft E. Different psychophysiological and behavioral responses elicited by frustration in pediatric bipolar disorder and severe mood dysregulation. Am J Psychiatry. 2007 Feb;164(2):309-17. doi: 10.1176/ajp.2007.164.2.309. PMID 17267795
- [Background] Rich BA, Schmajuk M, Perez-Edgar KE, Pine DS, Fox NA, Leibenluft E. The impact of reward, punishment, and frustration on attention in pediatric bipolar disorder. Biol Psychiatry. 2005 Oct 1;58(7):532-9. doi: 10.1016/j.biopsych.2005.01.006. Epub 2005 Jun 13. PMID 15953589
- [Background] Riem MM, Bakermans-Kranenburg MJ, Pieper S, Tops M, Boksem MA, Vermeiren RR, van Ijzendoorn MH, Rombouts SA. Oxytocin modulates amygdala, insula, and inferior frontal gyrus responses to infant crying: a randomized controlled trial. Biol Psychiatry. 2011 Aug 1;70(3):291-7. doi: 10.1016/j.biopsych.2011.02.006. Epub 2011 Apr 5. PMID 21470595
- [Background] Roca CA, Schmidt PJ, Altemus M, Deuster P, Danaceau MA, Putnam K, Rubinow DR. Differential menstrual cycle regulation of hypothalamic-pituitary-adrenal axis in women with premenstrual syndrome and controls. J Clin Endocrinol Metab. 2003 Jul;88(7):3057-63. doi: 10.1210/jc.2002-021570. PMID 12843143
- [Background] Roca CA, Schmidt PJ, Deuster PA, Danaceau MA, Altemus M, Putnam K, Chrousos GP, Nieman LK, Rubinow DR. Sex-related differences in stimulated hypothalamic-pituitary-adrenal axis during induced gonadal suppression. J Clin Endocrinol Metab. 2005 Jul;90(7):4224-31. doi: 10.1210/jc.2004-2525. Epub 2005 May 10. PMID 15886244
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397
- [Background] Rubin, D. B. (1987). Multiple Imputation for Nonresponse in Surveys. John Wiley & Sons.
- [Background] Saleh AA, Ginsburg KA, Duchon TA, Dorey LG, Hirata J, Alshameeri RS, Dombrowski MP, Mammen EF. Hormonal contraception and platelet function. Thromb Res. 1995 May 15;78(4):363-7. doi: 10.1016/0049-3848(95)91464-v. PMID 7631316
- [Background] Salum GA, Mogg K, Bradley BP, Stringaris A, Gadelha A, Pan PM, Rohde LA, Polanczyk GV, Manfro GG, Pine DS, Leibenluft E. Association between irritability and bias in attention orienting to threat in children and adolescents. J Child Psychol Psychiatry. 2017 May;58(5):595-602. doi: 10.1111/jcpp.12659. Epub 2016 Oct 26. PMID 27782299
- [Background] Sanchez LA, Moran C, Reyna R, Ochoa T, Boots LR, Azziz R. Adrenal progestogen and androgen production in 21-hydroxylase-deficient nonclassic adrenal hyperplasia is partially independent of adrenocorticotropic hormone stimulation. Fertil Steril. 2002 Apr;77(4):750-3. doi: 10.1016/s0015-0282(01)03236-8. PMID 11937128
- [Background] Sauer MV, Paulson RJ, Lobo RA. Reversing the natural decline in human fertility. An extended clinical trial of oocyte donation to women of advanced reproductive age. JAMA. 1992 Sep 9;268(10):1275-9. doi: 10.1001/jama.268.10.1275. PMID 1507373
- [Background] Savage J, Verhulst B, Copeland W, Althoff RR, Lichtenstein P, Roberson-Nay R. A genetically informed study of the longitudinal relation between irritability and anxious/depressed symptoms. J Am Acad Child Adolesc Psychiatry. 2015 May;54(5):377-84. doi: 10.1016/j.jaac.2015.02.010. Epub 2015 Feb 28. PMID 25901774
- [Background] Schiller CE, Johnson SL, Abate AC, Schmidt PJ, Rubinow DR. Reproductive Steroid Regulation of Mood and Behavior. Compr Physiol. 2016 Jun 13;6(3):1135-60. doi: 10.1002/cphy.c150014. PMID 27347888
- [Background] Schmidt PJ, Nieman LK, Danaceau MA, Adams LF, Rubinow DR. Differential behavioral effects of gonadal steroids in women with and in those without premenstrual syndrome. N Engl J Med. 1998 Jan 22;338(4):209-16. doi: 10.1056/NEJM199801223380401. PMID 9435325
- [Background] Schmidt PJ, Steinberg EM, Negro PP, Haq N, Gibson C, Rubinow DR. Pharmacologically induced hypogonadism and sexual function in healthy young women and men. Neuropsychopharmacology. 2009 Feb;34(3):565-76. doi: 10.1038/npp.2008.24. Epub 2008 Mar 19. PMID 18354393
- [Background] Scott LN, Stepp SD, Hallquist MN, Whalen DJ, Wright AGC, Pilkonis PA. Daily shame and hostile irritability in adolescent girls with borderline personality disorder symptoms. Personal Disord. 2015 Jan;6(1):53-63. doi: 10.1037/per0000107. PMID 25580673
- [Background] Scribner DR Jr, Walker JL. Low-grade endometrial stromal sarcoma preoperative treatment with Depo-Lupron and Megace. Gynecol Oncol. 1998 Dec;71(3):458-60. doi: 10.1006/gyno.1998.5174. PMID 9887250
- [Background] Simon JJ, Walther S, Fiebach CJ, Friederich HC, Stippich C, Weisbrod M, Kaiser S. Neural reward processing is modulated by approach- and avoidance-related personality traits. Neuroimage. 2010 Jan 15;49(2):1868-74. doi: 10.1016/j.neuroimage.2009.09.016. Epub 2009 Sep 18. PMID 19770056
- [Background] Smith SM, Jenkinson M, Woolrich MW, Beckmann CF, Behrens TE, Johansen-Berg H, Bannister PR, De Luca M, Drobnjak I, Flitney DE, Niazy RK, Saunders J, Vickers J, Zhang Y, De Stefano N, Brady JM, Matthews PM. Advances in functional and structural MR image analysis and implementation as FSL. Neuroimage. 2004;23 Suppl 1:S208-19. doi: 10.1016/j.neuroimage.2004.07.051. PMID 15501092
- [Background] Smoski MJ, Felder J, Bizzell J, Green SR, Ernst M, Lynch TR, Dichter GS. fMRI of alterations in reward selection, anticipation, and feedback in major depressive disorder. J Affect Disord. 2009 Nov;118(1-3):69-78. doi: 10.1016/j.jad.2009.01.034. Epub 2009 Mar 3. PMID 19261334
- [Background] Spinelli MG, Endicott J, Goetz RR, Segre LS. Reanalysis of efficacy of interpersonal psychotherapy for antepartum depression versus parenting education program: initial severity of depression as a predictor of treatment outcome. J Clin Psychiatry. 2016 Apr;77(4):535-40. doi: 10.4088/JCP.15m09787. PMID 27137422
- [Background] Stampfer MJ, Colditz GA, Willett WC, Manson JE, Rosner B, Speizer FE, Hennekens CH. Postmenopausal estrogen therapy and cardiovascular disease. Ten-year follow-up from the nurses' health study. N Engl J Med. 1991 Sep 12;325(11):756-62. doi: 10.1056/NEJM199109123251102. PMID 1870648
- [Background] Stefanick ML, Anderson GL, Margolis KL, Hendrix SL, Rodabough RJ, Paskett ED, Lane DS, Hubbell FA, Assaf AR, Sarto GE, Schenken RS, Yasmeen S, Lessin L, Chlebowski RT; WHI Investigators. Effects of conjugated equine estrogens on breast cancer and mammography screening in postmenopausal women with hysterectomy. JAMA. 2006 Apr 12;295(14):1647-57. doi: 10.1001/jama.295.14.1647. PMID 16609086
- [Background] Steinauer JE, Waetjen LE, Vittinghoff E, Subak LL, Hulley SB, Grady D, Lin F, Brown JS. Postmenopausal hormone therapy: does it cause incontinence? Obstet Gynecol. 2005 Nov;106(5 Pt 1):940-5. doi: 10.1097/01.AOG.0000180394.08406.15. PMID 16260510
- [Background] Steingold KA, Matt DW, DeZiegler D, Sealey JE, Fratkin M, Reznikov S. Comparison of transdermal to oral estradiol administration on hormonal and hepatic parameters in women with premature ovarian failure. J Clin Endocrinol Metab. 1991 Aug;73(2):275-80. doi: 10.1210/jcem-73-2-275. PMID 1906893
- [Background] Stoddard J, Tseng WL, Kim P, Chen G, Yi J, Donahue L, Brotman MA, Towbin KE, Pine DS, Leibenluft E. Association of Irritability and Anxiety With the Neural Mechanisms of Implicit Face Emotion Processing in Youths With Psychopathology. JAMA Psychiatry. 2017 Jan 1;74(1):95-103. doi: 10.1001/jamapsychiatry.2016.3282. PMID 27902832

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous OC
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Continuous OC
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.0 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-intervention to Intervention Endpoint in Weekly Average Binge-eating Frequency
Description: Binge eating frequency is based on a weekly diary of self-reported binge eating frequency. Participants were asked how many times during the past week they had a binge eating episode. Scores can range from 0 to infinity as frequency is self-reported as the number of binge eating episodes in the previous week. Higher scores indicate more episodes of binge eating. Change is defined as the average change in self-reported binge eating frequency from pre-intervention to intervention.
Time Frame: Pre-intervention (week 1) to intervention endpoint (week 12)
Population: Participants that started the study medication and completed the pre-intervention and intervention endpoints.
Measure: Mean (Standard Deviation); unit: episodes/week
Arm/Group | Continuous OC
Number analyzed (Participants) | 7
episodes/week | -0.43 (1.27)

2. Primary Outcome: Change From Pre-intervention to Intervention Endpoint in Binge Eating Sum Score
Description: Binge eating will be measured using the 8-item binge eating subscale of the Eating Pathology Symptoms Inventory (EPSI), which measures features of binge eating (e.g., consumption of large quantities of food, mindless eating) on a 5-point Likert scale from "never" to "very often." The EPSI scale is designed to assess behavior over the past 28 days. Items are summed for a scale score ranging from 0-32. Higher scores indicate more frequent experiences with binge eating behavior. Change is defined as the average change in the binge eating scale score from pre-intervention to intervention.
Time Frame: Pre-intervention (week 1) to intervention endpoint (week 12)
Population: Participants who started the study medication and completed the pre-intervention and intervention endpoints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous OC
Number analyzed (Participants) | 7
score on a scale | -6.60 (7.11)

3. Primary Outcome: Change From Pre-intervention to Intervention Endpoint in Nucleus Accumbens Signal Intensity in Response to Reward During the Monetary Incentive Delay Task (MIDT)
Description: Nucleus Accumbens (NAcc) reactivity to reward during the Monetary Incentive Delay (MIDT) task compared pre and post treatment. During MIDT task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when they see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared pre- and post-treatment.
Time Frame: Pre-intervention (week 1) to intervention endpoint (week 12)
Population: Participants who started the study medication and completed the pre-intervention and intervention endpoints. Due to technological error when saving data, one participant's endpoint MRI data was unusable.
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | Continuous OC
Number analyzed (Participants) | 6
percentage signal change | .0423 (.26)

4. Primary Outcome: Change From Pre-intervention to Intervention Endpoint in Dorsal Striatum Signal Intensity in Response to Reward During the Monetary Incentive Delay Task (MIDT)
Description: Dorsal striatum reactivity (defined as caudate signal intensity and putamen signal intensity) to reward during the Monetary Incentive Delay (MIDT) task compared pre and post treatment. During MIDT task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when they see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared pre- and post-treatment.
Time Frame: Pre-intervention (week 1) to intervention endpoint (week 12)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | Continuous OC
Number analyzed (Participants) | 6
percentage signal change
  Caudate | -.012 (.11)
  Putamen | .02 (.10)

5. Primary Outcome: Change From Pre-intervention to Intervention Endpoint in Prefrontal Cortex Signal Intensity in Response to Reward During the Monetary Incentive Delay Task (MIDT)
Description: Prefrontal cortex reactivity to reward during the Monetary Incentive Delay (MIDT) task compared pre and post treatment. During MIDT task, participants respond to "win" trials by pressing a button on a button box in the MRI as quickly as possible when they see a target. Reactivity is measured by examining participant's change in blood-oxygen-level dependent (BOLD) (i.e., measurement of oxygen level that is carried to neurons by red blood cells since areas of the brain that are thought to be more "active" or involved in certain tasks require more oxygen) in response to a stimulus of interest (win trials) versus non-stimulus (non-win trials). Percent signal change in BOLD activation between monetary reward versus non-reward is the outcome of interest. Percent signal change is then compared pre- and post-treatment.
Time Frame: Pre-intervention (week 1) to intervention endpoint (week 12)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | Continuous OC
Number analyzed (Participants) | 6
percentage signal change | .01 (.15)

6. Primary Outcome: Change From Pre-intervention to Intervention Endpoint in Delay Discounting Parameter k
Description: The Monetary Choice Questionnaire will be used to measure delay discounting. Participants will be asked to make a series of hypothetical choices between small, sooner (impulsive) vs. larger, later (self controlled) hypothetical monetary outcomes. k is a hyperbolic function with larger k values indicating more valuation of a larger delayed reward and smaller values indicating preference for more immediate, smaller rewards (more impulsivity). k can range from 0 to .25 with scores of .25 indicating complete valuation of the immediate reward and 0 indicating complete valuation of the larger, delayed reward. Change is defined as the average change in k from pre-intervention to intervention.
Time Frame: Pre-intervention (week 1) to intervention endpoint (week 12)
Population: Participants that started the study medication and completed the pre-intervention and intervention endpoints.
Measure: Mean (Standard Deviation); unit: k value
Arm/Group | Continuous OC
Number analyzed (Participants) | 7
k value | .01 (.013)

7. Secondary Outcome: Change From Pre-intervention to Intervention Endpoint in Self-reported Reward Sensitivity Subscale Score
Description: Sensitivity to Punishment/Sensitivity to Reward Questionnaire will be used to measure reward sensitivity. The reward sensitivity subscale will be used, which is rated on a true/false scale with scores ranging 0-24. Higher scores indicate more sensitivity to reward. Change is defined as the average change in reward sensitivity from pre-intervention to intervention.
Time Frame: Pre-intervention (week 1) to intervention endpoint (week 12)
Population: Participants that started the study medication and completed the pre-intervention and intervention endpoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous OC
Number analyzed (Participants) | 7
score on a scale | 1.60 (2.30)

8. Secondary Outcome: Change From Pre-intervention to Intervention Endpoint in Behavioral Inhibition Subscale Score
Description: The Behavioral Inhibition/Behavioral Activation questionnaire will be used to assess behavioural inhibition (BI). The minimum score on the BI subscale is 7, maximum 28. Greater scores indicate greater BI. Change is defined as the average change in BI from pre-intervention to intervention.
Time Frame: Pre-intervention (week 1) to intervention endpoint (week 12)
Population: Participants that started the study medication and completed the pre-intervention and intervention endpoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuous OC
Number analyzed (Participants) | 7
score on a scale | 1.43 (5.41)

ADVERSE EVENTS:
Time Frame: Adverse event data was tracked over a participant's time in the protocol (approximately 84 days).
Description: All unresolved adverse events were tracked by the investigator until the events were resolved, the subject was lost to follow-up, or the adverse event was otherwise explained.
Arm/Group | Continuous OC
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous OC (N=8)
Menstrual Bleeding (Reproductive system and breast disorders) | 4 (7)
Bloating (Endocrine disorders) | 2 (2)
Breast Tenderness (Reproductive system and breast disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Cramps (Reproductive system and breast disorders) | 3 (4) — Menstrual-type cramps
Irritability (Psychiatric disorders) | 2 (2)
Spotting (Reproductive system and breast disorders) | 8 (14)
Lethargic (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (4)
Low Mood (Psychiatric disorders) | 1 (1)
Drowsiness (General disorders) | 2 (2)
Mood Change (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Insomnia (General disorders) | 1 (1)
Decreased Overeating (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to the inability to recruit eligible participants therefore only a very small number of participants have available data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04278755/Prot_SAP_000.pdf